CLINICAL TRIAL: NCT00365313
Title: A Phase 3 Double Blinded, Randomized, Placebo Controlled Trial of Proton Pump Inhibitor for the Prevention of Recurrent Ulcer Bleeding in Patients Receiving a COX-2 Inhibitor
Brief Title: Preventing Recurrent Ulcer Bleeding in Arthritis Patients Using Esomeprazole Plus Celecoxib
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7NB study
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2006-10-27 (Estimated); Status verified 2006-10

CONDITIONS: Arthritis; Bleeding Ulcer
Keywords: celecoxib; oesomeprazole; arthritis; ulcer bleeding
MeSH Terms: conditions — Arthritis | interventions — Celecoxib; Esomeprazole

INTERVENTIONS:
Drug: celecoxib, esomeprazole

SUMMARY:
The purpose of this study is to compare the effect of Esomeparzole with Placebo in the Prevention of Recurrent Ulcer Bleeding in Patients Receiving a COX-2 Inhibitor

DETAILED DESCRIPTION:
Among patients with previous ulcer bleeding, neither nonsteroidal anti-inflammatory drugs (NSAIDs) plus a proton pump inhibitor (PPI) nor a cyclooxygenase (COX)-2 inhibitor adequately prevents recurrent ulcer bleeding.

The aim is to investigate whether adding a PPI to a COX-2 inhibitor is superior to a COX-2 inhibitor alone for the prevention of recurrent ulcer bleeding in high-risk patients.

Patients with arthritis who presented with NSAID-induced ulcer bleeding were eligible if they had healed ulcers on follow-up endoscopy; were H. pylori negative or eradicated; and required regular NSAIDs. After the ulcers had healed, all patients received celecoxib 200 mg b.i.d. They were randomly assigned to esomeprazole 20 mg b.i.d. or its placebo for 12 months. The primary endpoint was recurrent ulcer bleeding.

Results Intention-to-treat analysis included 273 patients (137 received esomeprazole and 136 received placebo). Recurrent ulcer bleeding occurred in none receiving esomeprazole and 8 patients receiving placebo. The 12-month cumulative incidence of recurrent bleeding was 0% in the esomeprazole group and 8.9% in the placebo group (difference, 8.9 percentage points; 95% confidence interval for the difference, 4.1 to 13.7; P=0.0004). During follow-up, 16.1% of patients in the esomeprazole group and 15.4% in the placebo group used low-dose aspirin. Among patients who did not use aspirin, the cumulative incidence of recurrent ulcer bleeding was 0% in the esomeprazole group and 7.1% in the placebo group (difference, 7.1 percentage points; 95% confidence interval, 2.4 to 11.8; P=0.004).

Conclusion Among patients with arthritis who have previous NSAID-induced ulcer bleeding, adding a PPI to a COX-2 inhibitor is superior to a COX-2 inhibitor alone for the prevention of recurrent ulcer bleeding.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were ulcer healing confirmed by follow-up endoscopy, a negative test for Helicobacter pylori or successful eradication of Helicobacter pylori based on histology, and anticipated regular use of NSAIDs for the duration of the trial. The exclusion criteria were concomitant use of low-dose aspirin, anticoagulants or corticosteroids; a history of gastric or duodenal surgery other than a patch repair; the presence of erosive esophagitis, gastric outlet obstruction, renal failure (defined by a serum creatinine level of more than 2.26 mg per deciliter), terminal illness, or cancer.

Exclusion Criteria:

* The exclusion criteria were concomitant use of low-dose aspirin, anticoagulants or corticosteroids; a history of gastric or duodenal surgery other than a patch repair; the presence of erosive esophagitis, gastric outlet obstruction, renal failure (defined by a serum creatinine level of more than 2.26 mg per deciliter), terminal illness, or cancer.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273
Dates: Start 2002-08; Study Completion 2005-06

PRIMARY OUTCOMES:
ulcer rebleeding over period of 13 months

SECONDARY OUTCOMES:
stroke or cardio-vascular events

CONTACTS AND LOCATIONS:
Overall Officials: Francis K Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Hong Kong, China

REFERENCES:
- [Derived] Chan FK, Wong VW, Suen BY, Wu JC, Ching JY, Hung LC, Hui AJ, Leung VK, Lee VW, Lai LH, Wong GL, Chow DK, To KF, Leung WK, Chiu PW, Lee YT, Lau JY, Chan HL, Ng EK, Sung JJ. Combination of a cyclo-oxygenase-2 inhibitor and a proton-pump inhibitor for prevention of recurrent ulcer bleeding in patients at very high risk: a double-blind, randomised trial. Lancet. 2007 May 12;369(9573):1621-6. doi: 10.1016/S0140-6736(07)60749-1. PMID 17499604